CLINICAL TRIAL: NCT00142948
Title: Heroin Addiction Treatment: Naltrexone and Adrenergic Agents
Brief Title: Naltrexone and Adrenergic Agents to Reduce Heroin Use in Heroin Addicts
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Thomas R. Kosten, MD, Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIDA-18863; R01DA018863 (NIH); DPMC
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Last update posted 2012-10-24 (Estimated); Status verified 2012-10

CONDITIONS: Heroin Dependence
Keywords: Heroin Abuse; Heroin Addiction
MeSH Terms: conditions — Heroin Dependence | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Naltrexone (Experimental): Naltrexone Oral 50 mgs daily
  Interventions: Drug: Naltrexone
- Placebo (Placebo Comparator): 1 to 1 comparison of Naltrexone to placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Naltrexone — naltrexone
  Arms: Naltrexone
Drug: Placebo — placebo
  Arms: Placebo

SUMMARY:
Naltrexone is a medication that is currently used to treat drug and alcohol addiction. Guanfacine is a medication that is currently used to manage the withdrawal symptoms in individuals undergoing opioid detoxification. A combination of these two medications may be beneficial in reducing heroin use in individuals addicted to heroin. This study will evaluate the effectiveness of naltrexone and guanfacine, alone and in combination, at reducing heroin use in heroin addicts.

DETAILED DESCRIPTION:
Heroin addiction is a serious health problem with no available medical treatment for preventing relapse. Naltrexone is a medication that is currently used to treat substance addiction. It acts by blocking the "high" feeling produced by drugs and alcohol. Guanfacine, an antihypertensive medication, is currently used to manage the withdrawal symptoms in individuals undergoing opioid detoxification. While each of these medications is useful in the treatment of heroin addiction, a combination of the two drugs may be more effective than either medication alone. The purpose of this study is to compare the effectiveness of naltrexone, guanfacine, and a combination of naltrexone and guanfacine at reducing drug relapse in heroin addicts.

This study will enroll individuals addicted to heroin who have completed a prior detoxification program at one of two addiction treatment hospitals in St. Petersburg, Russian Federation. Upon completing the detoxification program of 7-14 days, participants will have a period of inpatient rehabilitation. During this 3- to 4-week inpatient stabilization period, patients will be screened for study participation. Once stabilized, participants will begin the 6-month treatment phase of the study. During this phase, they will be randomly assigned to receive one of the following drug combinations on a daily basis: 50 mg of naltrexone and guanfacine placebo; 1.0 mg of guanfacine and naltrexone placebo; 50 mg of naltrexone and 1.0 mg of guanfacine; or naltrexone placebo and guanfacine placebo. All participants will have a designated family member who will be responsible for supervising medication compliance. Study visits will occur twice monthly. Participants will receive clinical management and medication compliance counseling at each visit; family members will also take part in the counseling sessions. Outcome measurements will include drug relapse, medication adherence, withdrawal symptoms, HIV risk factors, and psychiatric symptoms. Follow-up evaluations will occur 3 and 6 months following the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Current primary diagnosis of heroin dependence, for at least 1 year prior to study entry
* High school graduate or higher education level
* Abstinence from drugs and alcohol for at least 1 week prior to study entry
* Negative urine and breathalyzer tests for alcohol and drugs
* No evidence of opioid dependence following narcan challenge
* At least one relative willing to participate in treatment, monitor administration of medications, assist in follow-up, and provide outcome data
* Stable address within St. Petersburg or nearest districts of Leningrad Region
* Able to provide a home telephone number where the participant may be reached
* If female, willing to use effective contraception throughout the study

Exclusion Criteria:

* Low blood pressure, as determined by sitting blood pressure less than 90/50 mm Hg
* Clinically significant cognitive impairment, schizophrenia, paranoid disorder, bipolar disorder, or seizure disorder
* Advanced brain, heart, kidney, or liver disease
* Active tuberculosis
* Current febrile illness
* AIDS-defining illness
* Significant laboratory abnormality, including severe anemia, unstable diabetes, or liver function tests greater than three times above normal
* Pending legal issues that may entail a jail stay during the study
* Currently participating in another treatment study
* Currently participating in another substance abuse program
* Current use of a psychotropic medication
* Pregnant
* Pulse rate less than 50 bpm

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 301 (Actual)
Dates: Start 2006-02; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Heroin relapse | duration of study

SECONDARY OUTCOMES:
HIV risk factors | baseline
Psychiatric symptoms (measured at Month 6, and the 3- and 6-month follow-up evaluations) | months 6 and the 3- and 6-month follow-up evaluations
Adherence to medication | duration of study
Heroin withdrawal symptoms | Month 6, and 3- and 6-month followup

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R. Kosten, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Saint Petersburg Pavlov State Medical University, Saint Petersburg, Russia